CLINICAL TRIAL: NCT02652624
Title: A Phase 3, Randomized, Open Label Study to Evaluate the Safety and Efficacy of Switching to a Fixed Dose Combination (FDC) of GS-9883/Emtricitabine/Tenofovir Alafenamide (GS-9883/F/TAF) From Elvitegravir/Cobicistat/Emtricitabine/ Tenofovir Alafenamide (E/C/F/TAF), Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Disoproxil Fumarate (E/C/F/TDF) or Atazanavir + Ritonavir + Emtricitabine/Tenofovir Disoproxil Fumarate (ATV+RTV+FTC/TDF) in Virologically Suppressed HIV-1 Infected Women
Brief Title: Safety and Efficacy of Switching to a FDC of B/F/TAF From E/C/F/TAF, E/C/F/TDF, or ATV+RTV+FTC/TDF in Virologically Suppressed HIV-1 Infected Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-380-1961
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2019-11

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Atazanavir Sulfate; Ritonavir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- B/F/TAF (Experimental): Participants will switch to B/F/TAF FDC and receive treatment for 48 weeks.
  Interventions: Drug: B/F/TAF
- Baseline Regimen (Active Comparator): Participants will remain on their baseline regimen of E/C/F/TAF, E/C/F/TDF, or ATV+RTV+FTC/TDF for 48 weeks.
  Interventions: Drug: E/C/F/TAF; Drug: E/C/F/TDF; Drug: ATV; Drug: RTV; Drug: FTC/TDF
- Extension Phase (Experimental): Following Week 48, participants in countries where B/F/TAF is not available may have the option to receive B/F/TAF for up to 48 additional weeks.
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: E/C/F/TAF — 150/150/200/10 mg FDC tablet administered orally once daily with food
  Other Names: Genvoya®
  Arms: Baseline Regimen
Drug: E/C/F/TDF — 150/150/200/300 mg FDC administered orally once daily with food
  Other Names: Stribild®
  Arms: Baseline Regimen
Drug: ATV — ATV 300 mg capsules administered orally once daily with food
  Other Names: Reyataz®
  Arms: Baseline Regimen
Drug: RTV — RTV 100 mg tablets administered orally once daily with food
  Other Names: Norvir®
  Arms: Baseline Regimen
Drug: FTC/TDF — 200/300 mg tablet administered orally once daily with food
  Other Names: Truvada®
  Arms: Baseline Regimen
Drug: B/F/TAF — 50/200/25 mg FDC tablet administered orally once daily without regard to food
  Other Names: Biktarvy®
  Arms: B/F/TAF; Extension Phase

SUMMARY:
The primary objective of this study is to evaluate the efficacy of switching to a fixed-dose combination (FDC) of bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) versus continuing on a regimen consisting of elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF), elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (E/C/F/TDF), or atazanavir (ATV) + ritonavir (RTV) + emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) in virologically suppressed HIV-1 infected women.

ELIGIBILITY:
Key Inclusion Criteria

Medically stable HIV-1 infected women who meet the following criteria:

* Completion of the Week 48 open-label extension (OLE) visit or any post Week 48 OLE visits in Gilead-sponsored study GS-US-236-0128, or Completion of the Week 96 visit or any post Week 96 visits in Gilead-sponsored study GS-US-292-0109 or completion of the Week 144 visit or any post Week 144 visits in Gilead sponsored studies GS-US-292-0104 or GS-US-292-0111.
* Currently on a stable antiretroviral regimen consisting of E/C/F/TAF, E/C/F/TDF, or ATV+RTV+FTC/TDF continuously for ≥ 12 consecutive weeks preceding the Screening visit
* Documented plasma HIV-1 RNA levels < 50 copies/mL for ≥ 12 weeks preceding the Screening visit. After reaching HIV-1 RNA < 50 copies/mL, single values of HIV-1 RNA

  ≥ 50 copies/mL followed by re-suppression to < 50 copies/mL is allowed
* HIV-1 RNA <50 copies/mL at screening
* Estimated glomerular filtration rate (eGFR) ≥ 50 mL/min (≥ 0.83 mL/sec) according to the Cockcroft-Gault formula at the Screening visit

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2017-10-09 (Actual); Study Completion 2018-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (46):
- United States (25):
  - Stamford, Connecticut
  - Washington D.C., District of Columbia
  - Fort Lauderdale, Florida
  - Ft. Pierce, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Macon, Georgia
  - Savannah, Georgia
  - Springfield, Massachusetts
  - St Louis, Missouri
  - Newark, New Jersey
  - Great Neck, New York
  - The Bronx, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Huntersville, North Carolina
  - Bellaire, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Harlingen, Texas
  - Houston, Texas
- Santo Domingo, Dominican Republic
- San Juan, Puerto Rico
- Russia (14):
  - Barnaul
  - Irkutsk
  - Khabarovsk
  - Krasnodar
  - Krasnoyarsk
  - Lipetsk
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg
  - Saint-Petersberg
  - Volgograd
  - Voronezh
  - Yekaterinburg
  - Коltsovo
- Thailand (4):
  - Bangkok
  - Chiang Mai
  - Khon Kaen
  - Nonthaburi
- Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Derived] Avihingsanon A, Chetchotisakd P, Kiertiburanakul S, Ratanasuwan W, Siripassorn K, Supparatpinyo K, Martin H, Wang H, Wong T, Wang HY. Efficacy and safety of switching to bictegravir, emtricitabine, and tenofovir alafenamide in virologically suppressed Asian adults living with HIV: A pooled analysis from three international phase III randomized trials. HIV Med. 2023 Mar;24(3):290-300. doi: 10.1111/hiv.13386. Epub 2022 Aug 17. PMID 36912172
- [Derived] Kityo C, Hagins D, Koenig E, Avihingsanon A, Chetchotisakd P, Supparatpinyo K, Gankina N, Pokrovsky V, Voronin E, Stephens JL, DeJesus E, Wang H, Acosta RK, Cao H, Quirk E, Martin H, Makadzange T. Switching to Fixed-Dose Bictegravir, Emtricitabine, and Tenofovir Alafenamide (B/F/TAF) in Virologically Suppressed HIV-1 Infected Women: A Randomized, Open-Label, Multicenter, Active-Controlled, Phase 3, Noninferiority Trial. J Acquir Immune Defic Syndr. 2019 Nov 1;82(3):321-328. doi: 10.1097/QAI.0000000000002137. PMID 31609930

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Russian Federation, Thailand, Dominican Republic, and Uganda. The first participant was screened on 19 February 2016. The last study visit occurred on 26 November 2018.
Pre-assignment Details: 491 participants were screened.
Groups:
- B/F/TAF: Randomized Phase: Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) (50/200/25 mg) fixed-dose combination (FDC) tablet once daily for at least 48 weeks, without regard to food.
  Extension Phase: After Week 48, participants in countries where B/F/TAF was not available were given the option to receive B/F/TAF (50/200/25 mg) FDC tablet once daily for up to 48 additional weeks, or until the product became accessible to participants through an access program, or until Gilead elected to discontinue the study in that country, whichever occurred first.
- Stay on Baseline Regimen (SBR): Randomized Phase: Participants remained on their baseline regimen of elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) (150/150/200/10 mg) tablet, elvitegravir/cobicistat/emtricitabine/tenofovir disoproxil fumarate (E/C/F/TDF) (150/150/200/300 mg) tablet, or atazanavir (ATV) 300 mg capsule + ritonavir (RTV) 100 mg tablet + emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) (200/300 mg) tablet for at least 48 weeks with food.
  Extension Phase: After Week 48, participants in countries where B/F/TAF was not available were given the option to receive B/F/TAF (50/200/25 mg) FDC tablet once daily for up to 48 additional weeks, or until the product became accessible to participants through an access program, or until Gilead elected to discontinue the study in that country, whichever occurred first.
Period: Randomized Phase
Arm/Group | B/F/TAF | Stay on Baseline Regimen (SBR)
Started | 234 | 236
Completed | 231 | 231
Not Completed | 3 | 5
Not completed — Pregnancy | 3 | 1
Not completed — Investigator's Discretion | 0 | 2
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Extension Phase
Arm/Group | B/F/TAF | Stay on Baseline Regimen (SBR)
Started | 231 | 228 (3 participants completed the Randomized Phase, but did not enter the Extension Phase.)
Completed | 227 | 224
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 3 | 1
Not completed — Pregnancy | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrew Consent | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Groups:
- B/F/TAF: B/F/TAF (50/200/25 mg) FDC tablet once daily without regard to food for 48 weeks.
- Stay on Baseline Regimen: Participants remained on their baseline regimen of E/C/F/TAF (150/150/200/10 mg) tablet, E/C/F/TDF (150/150/200/300 mg) tablet, or ATV 300 mg capsule + RTV 100 mg tablet + FTC/TDF (200/300 mg) tablet for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | B/F/TAF | Stay on Baseline Regimen | Total
Number analyzed (Participants) | 234 | 236 | 470
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (9.5) | 40 (9.1) | 40 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 234 | 236 | 470
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 38 | 74
  Not Hispanic or Latino | 198 | 198 | 396
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 48 | 54 | 102
  Black | 91 | 83 | 174
  White | 66 | 67 | 133
  Other | 29 | 32 | 61
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 36 | 72
  Dominican Republic | 28 | 30 | 58
  Uganda | 65 | 62 | 127
  Thailand | 47 | 54 | 101
  Russia | 58 | 54 | 112
HIV-1 RNA Category [Count of Participants; unit: Participants]
  < 50 copies/mL | 234 | 233 | 467
  ≥ 50 copies/mL | 0 | 3 | 3
CD4 Cell Count [Mean (Standard Deviation); unit: cells/µL] | 712 (268.1) | 738 (268.4) | 725 (268.3)
CD4 Cell Count Category [Count of Participants; unit: Participants]
  ≥ 50 to < 200 cells/µL | 1 | 1 | 2
  ≥ 200 to < 350 cells/µL | 10 | 9 | 19
  ≥ 350 to < 500 cells/µL | 33 | 25 | 58
  ≥ 500 cells/µL | 190 | 201 | 391
Prior Antiretroviral (ARV) Regimen [Count of Participants; unit: Participants]
  E/C/F/TAF | 124 | 125 | 249
  E/C/F/TDF | 99 | 98 | 197
  RTV + ATV + FTC/TDF | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA ≥ 50 Copies/mL at Week 48 as Determined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: The Full Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | Stay on Baseline Regimen
Number analyzed (Participants) | 234 | 236
percentage of participants | 1.7 | 1.7
Statistical Analysis 1: Comparison: B/F/TAF vs Stay on Baseline Regimen; The null hypothesis was that the percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48 in the B/F/TAF group was at least 4% higher than the rate in the SBR group; the alternative hypothesis was that the percentage of participants with HIV-1 RNA ≥ 50 copies/mL in the B/F/TAF group was less than 4% higher than that in the SBR group; Test type: Non-Inferiority — A sample size of 470 participants (~235 participants per treatment group) would provide at least 87% power to detect a non-inferiority margin of 4% difference in the percentage of participants with HIV-1 RNA ≥ 50 copies/mL at Week 48 between the 2 treatment groups. This was based on the assumptions that both treatment groups have 2% of participants with HIV-1 RNA ≥ 50 copies/mL (based on Gilead Genvoya and Stribild studies) and that the significance level of the test is at a 1-sided 0.025 level; Difference in percentages = 0.0, 95.001% CI 2-sided [-2.9 to 2.9] — The difference in percentages between treatment groups and their 95.001% confidence intervals (CI) were calculated based on an unconditional exact method using 2 inverted 1-sided tests
Statistical Analysis 2: Comparison: B/F/TAF vs Stay on Baseline Regimen; Test type: Superiority; p = 1.00, Fisher Exact

2. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 as Determined by the US FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF | Stay on Baseline Regimen
Number analyzed (Participants) | 234 | 236
percentage of participants | 95.7 | 95.3
Statistical Analysis 1: Comparison: B/F/TAF vs Stay on Baseline Regimen; Test type: Non-Inferiority — The non-inferiority of B/F/TAF would be established if the lower bound of the 2-sided 95.001% CI of the difference between the treatment groups (B/F/TAF group - SBR group) in the percentage of participants with HIV-1 RNA < 50 copies/mL is greater than -10%; Difference in percentages = 0.4, 95.001% CI 2-sided [-3.7 to 4.5] — The difference in percentages between treatment groups and their 95.001% CIs were calculated based on an unconditional exact method using 2 inverted 1-sided tests
Statistical Analysis 2: Comparison: B/F/TAF vs Stay on Baseline Regimen; Test type: Superiority; p = 1.00, Fisher Exact

3. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | B/F/TAF | Stay on Baseline Regimen
Number analyzed (Participants) | 225 | 225
cells/µL | 29 (159.4) | 26 (170.3)
Statistical Analysis 1: Comparison: B/F/TAF vs Stay on Baseline Regimen; Test type: Other; p = 0.84, ANOVA; Difference in least square means = 3, 95% CI 2-sided [-27 to 34] — Difference in least squares means and its 95% CI were from ANOVA model with treatment group as a fixed effect in the model

ADVERSE EVENTS:
Time Frame: First dose date to last dose date (maximum duration: 128.4 weeks) plus 30 days
Description: The Safety Analysis Set included participants who were randomized and received at least 1 dose of study drug.
Groups:
- B/F/TAF (Randomized Phase): Adverse events reported occurred during the Randomized Phase in participants from the B/F/TAF group, who received B/F/TAF (50/200/25 mg) FDC tablet once daily without regard to food for 48 weeks.
- Stay on Baseline Regimen (Randomized Phase): Adverse events reported occurred during the Randomized Phase in participants from the SBR group, who remained on their baseline regimen of E/C/F/TAF (150/150/200/10 mg) tablet, E/C/F/TDF (150/150/200/300 mg) tablet, or ATV 300 mg capsule + RTV 100 mg tablet + FTC/TDF (200/300 mg) tablet for 48 weeks.
- Extension Phase B/F/TAF From B/F/TAF: Adverse events reported occurred during the Extension Phase in participants who enrolled into the Extension Phase from the B/F/TAF group and received B/F/TAF (50/200/25 mg) FDC tablet for up to 48 additional weeks, or until the product became accessible to participants through an access program, or until Gilead elected to discontinue the study in that country, whichever occurred first.
- Extension Phase B/F/TAF From Stay on Baseline Regimen: Adverse events reported occurred during the Extension Phase in participants who enrolled into the Extension Phase from the SBR group and received B/F/TAF (50/200/25 mg) FDC tablet for up to 48 additional weeks, or until the product became accessible to participants through an access program, or until Gilead elected to discontinue the study in that country, whichever occurred first.
Arm/Group | B/F/TAF (Randomized Phase) | Stay on Baseline Regimen (Randomized Phase) | Extension Phase B/F/TAF From B/F/TAF | Extension Phase B/F/TAF From Stay on Baseline Regimen
All-Cause Mortality (participants affected / at risk) | 0/234 | 0/236 | 0/231 | 1/228
Serious Adverse Events (participants affected / at risk) | 7/234 | 9/236 | 8/231 | 10/228
Other Adverse Events (participants affected / at risk) | 61/234 | 47/236 | 52/231 | 41/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF (Randomized Phase) (N=234) | Stay on Baseline Regimen (Randomized Phase) (N=236) | Extension Phase B/F/TAF From B/F/TAF (N=231) | Extension Phase B/F/TAF From Stay on Baseline Regimen (N=228)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Urachal abnormality (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Abdominal wall abscess (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0
Malaria (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1 | 0
Salpingo-oophoritis (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Device issue (Product Issues) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Substance use (Social circumstances) | 0 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF (Randomized Phase) (N=234) | Stay on Baseline Regimen (Randomized Phase) (N=236) | Extension Phase B/F/TAF From B/F/TAF (N=231) | Extension Phase B/F/TAF From Stay on Baseline Regimen (N=228)
Nasopharyngitis (Infections and infestations) | 18 | 15 | 19 | 13
Upper respiratory tract infection (Infections and infestations) | 15 | 14 | 19 | 15
Urinary tract infection (Infections and infestations) | 16 | 4 | 8 | 5
Vulvovaginal candidiasis (Infections and infestations) | 12 | 9 | 9 | 9
Headache (Nervous system disorders) | 12 | 13 | 13 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (5):
  • Study Protocol: Original (2015-11-20): https://cdn.clinicaltrials.gov/large-docs/24/NCT02652624/Prot_000.pdf
  • Study Protocol: Amendment 1 (2016-06-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT02652624/Prot_001.pdf
  • Study Protocol: Amendment 2 (2016-11-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT02652624/Prot_002.pdf
  • Statistical Analysis Plan: Week 48 Statistical Analysis Plan (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT02652624/SAP_003.pdf
  • Statistical Analysis Plan: Final Statistical Analysis Plan (2018-12-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT02652624/SAP_004.pdf